CLINICAL TRIAL: NCT03719105
Title: Pilot Study Using Induction Chemo-immunotherapy Followed by Consolidation With Reduced Toxicity Conditioning and Allogenic Stem Cell Transplant in Advanced Stage Mature Non-anaplastic T-Cell or NK Lymphoma/Leukemia in Children, Adolescents and Young Adults; A NK/T-Cell Lymphoma/Leukemia Consortium Study
Brief Title: Chemoimmunotherapy and Allogeneic Stem Cell Transplant for NK T-cell Leukemia/Lymphoma
Status: Recruiting | Phase: Early Phase 1 | Type: Interventional
Sponsor: New York Medical College (Other)
Collaborators: University of Alabama at Birmingham (Other)
Responsible Party: Principal Investigator, Mitchell Cairo, Executive Vice-Chair, New York Medical College
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: NYMC 575
Record Dates: First submitted 2018-10-23; First posted 2018-10-25 (Actual); Last update posted 2025-08-08 (Actual); Status verified 2025-08

CONDITIONS: NK-Cell Lymphoma; NK-Cell Leukemia; Peripheral T Cell Lymphoma
MeSH Terms: conditions — Leukemia, Large Granular Lymphocytic; Lymphoma, T-Cell, Peripheral | interventions — Methotrexate; Ifosfamide; Dexamethasone; Etoposide; calaspargase pegol; Cyclophosphamide; Doxorubicin; Prednisone; Brentuximab Vedotin

STUDY DESIGN:
Intervention Model Description: Cohort 1 and 2 will be based on initial diagnosis.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Cohort 1 (Experimental): Patients with aggressive NK cell leukemia or stage III or IV extranodal NK/T-cell lymphoma, nasal type.
  Chemotherapy Regimen:
  mSMILE: Methotrexate Day 1, Ifosfamide Days 2-4, Dexamethasone Days 2-4, Etoposide Days 2-4, calaspargase pegol Day 8. For patients in CR and no available allogeneic SCT can receive up to 2 additional cycles of mSMILE.
  Pembrolizumab: For patients in PR/MR/NR/PD after 2 cycles of mSMILE.
  Allogeneic Stem Cell Transplant if donor available and not in PD.
  Interventions: Drug: Methotrexate; Drug: Ifosfamide; Drug: Dexamethasone; Drug: Etoposide; Drug: calaspargase pegol
- Cohort 2 (Experimental): Patients with stage III or IV peripheral T-cell lymphoma-NOS, angioimmunoblastic T-cell lymphoma, hepatosplenic T-cell lymphoma, or enteropathy-associated T-cell lymphoma (other histologies will be considered after case-by-case discussion with Study Chairs and Executive Vice-Chairs).
  Chemotherapy Regimen:
  Cycle 1 & 2: Pralatrexate Days 1, 8, and 15, cyclophosphamide Day 1, DOXOrubicin Day 1, predniSONE days 1-5 Cycle 3 & 5: Brentuximab vedotin Day 1, cyclophosphamide Day 1, DOXOrubicin Day 1, predniSONE days 1-5 Cycle 4 & 6: Pralatrexate Days 1, 8, and 15, cyclophosphamide Day 1, DOXOrubicin Day 1, predniSONE days 1-5 Allogeneic Stem Cell Transplant if donor available and not in PD.
  Interventions: Drug: pralatraxate,; Drug: cyclophosphamide; Drug: Doxorubicin; Drug: Prednisone; Drug: Brentuximab Vedotin

INTERVENTIONS:
Drug: Methotrexate — Patients will receive methotrexate as part of chemoimmunotherapy regemin followed by allogeneic stem cell transplant.
  Arms: Cohort 1
Drug: pralatraxate, — Patients will receive pralaxtraxate as part of chemoimmunotherapy regimen followed by allogeneic stem cell transplant.
  Arms: Cohort 2
Drug: Ifosfamide — Patients will receive Ifsofamide as part of chemoimmunotherapy regimen followed by allogeneic stem cell transplant.
  Arms: Cohort 1
Drug: Dexamethasone — Patients will receive dexamethasone as part of chemoimmunotherapy regimen followed by allogeneic stem cell transplant.
  Arms: Cohort 1
Drug: Etoposide — Patients will receive etoposide as part of chemoimmunotherapy regimen followed by allogeneic stem cell transplant.
  Arms: Cohort 1
Drug: calaspargase pegol — Patients will receive pegaspargase as part of chemoimmunotherapy regimen followed by allogeneic stem cell transplant.
  Arms: Cohort 1
Drug: cyclophosphamide — Patients will receive cyclophosphamide as part of chemoimmunotherapy regimen followed by allogeneic stem cell transplant.
  Arms: Cohort 2
Drug: Doxorubicin — Patients will receive doxorubicin as part of chemoimmunotherapy regimen followed by allogeneic stem cell transplant.
  Arms: Cohort 2
Drug: Prednisone — Patients will receive prednisone as part of chemoimmunotherapy regimen followed by allogeneic stem cell transplant.
  Arms: Cohort 2
Drug: Brentuximab Vedotin — Patients will receive brentuximab vedotin as part of chemoimmunotherapy regimen followed by allogeneic stem cell transplant.
  Arms: Cohort 2

SUMMARY:
Patients are in 2 cohorts:

Cohort 1: dexamethasone, methotrexate, ifosfamide, pegaspargase, and etoposide (modified SMILE) chemotherapy regimen alone and pembrolizumab in children, adolescents, and young adults with advanced stage NK lymphoma and leukemia Cohort 2: combining pralatrexate (PRX) (Cycles 1, 2, 4, 6) and brentuximab vedotin (BV) (Cycles 3, 5) to cyclophosphamide, doxorubicin, and prednisone in children, adolescent, and young adults with advanced peripheral T-cell lymphoma (non-anaplastic large cell lymphoma or non-NK lymphoma/leukemia) .

Both groups proceed to allogeneic stem cell transplant with disease response.

ELIGIBILITY:
Inclusion Criteria:

* Patients must weigh at least 10 kilograms at the time of the study enrollment.
* Diagnosis

Newly diagnosed patients with histologically proven mature T- and NK- cell neoplasms:

COHORT 1

* Aggressive NK cell leukemia (ICD-O code 9948/3)
* Extranodal NK/T-cell lymphoma, nasal type (ICD-O code 9719/3) COHORT 2
* Enteropathy-associated T-cell lymphoma (ICD-O code 9717/3)
* Hepatosplenic T-cell lymphoma (ICD-O code 9716/3)
* Peripheral T-cell lymphoma, non-otherwise specified (ICD-O code 9702/3)
* Angioimmunoblastic T-cell lymphoma (ICD-O code 9705/3)
* Other mature T- and NK-cell neoplasm histologies will considered after case-by-case discussion with Study Chairs and executive Vice-Chair Patients with lymphoma must have stage III or IV disease (See Appendix III for Staging).

  * Organ Function Requirements

Adequate liver function defined as:

* Total bilirubin ≤ 1.5 x upper limit of normal (ULN) for age.
* ALT (SGPT) < 3 x ULN for age.

Adequate cardiac function defined as:

* Shortening fraction of ≥ 27% by echocardiogram, or
* Ejection fraction of ≥ 50% by radionuclide angiogram.

Adequate pulmonary function defined as:

• Patients with a history of pulmonary dysfunction must have no evidence of dyspnea at rest, no exercise intolerance due to pulmonary insufficiency, and a pulse oximetry > 92% while breathing room air unless current dysfunction is due to the lymphoma, in which case the patient is eligible.

Exclusion Criteria:

* Alk+ or Alk- Anaplastic Large Cell Lymphoma (ALCL)
* Patients with active CNS disease.
* Patients with stage I or stage II disease (See Appendix III for Staging).
* Patients who have received any prior cytotoxic chemotherapy for the current diagnosis of NHL.
* Previous steroid treatment and/or radiation treatment are not allowed unless they are used for emergency management. Patients who have received emergency irradiation and/or steroid therapy will be eligible only if started on protocol therapy not more than one week from the start of radiotherapy or steroids.
* Female patients who are pregnant. Pregnancy tests must be obtained in girls who are post menarchal.
* Lactating females, unless they have agreed not to breastfeed their infants.
* Patients with Down syndrome.
* Patients taking CYP3A4 substrates with narrow therapeutic indices. Patients (COHORT 2 ONLY) chronically receiving medications known to be metabolized by CYP3A4 and with narrow therapeutic indices (See Appendix V). The topical use of these medications (if applicable) is allowed.
* Patients taking CYP3A4 inhibitors. Patients (COHORT 2 ONLY) chronically receiving drugs that are known potent CYP3A4 inhibitors within 7 days prior to study enrollment (See Appendix V). The topical use of these medications (if applicable) is allowed.
* Patients taking CYP3A4 inducers. Patients (COHORT 2 ONLY) chronically receiving drugs that are known potent CYP3A4 inducers within 12 days prior to study enrollment (See Appendix V).

Ages: 1 Year to 31 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 40 (Estimated)
Dates: Start 2019-03-01 (Actual); Primary Completion 2027-12-31 (Estimated); Study Completion 2028-12-31 (Estimated)

PRIMARY OUTCOMES:
overall response rate | 1 year
  to assess overall response rate following chemoimmunotherapy induction therapy

SECONDARY OUTCOMES:
event free survival | 2 year
  to determine the event free survival after induction chemoimmunotherapy and allogeneic stem cell transplantation

CONTACTS AND LOCATIONS:
Overall Officials: Mitchell Cairo, MD, Study Director — New York Medical College
Locations (6):
- United States (6):
  - University of Alabama, Birmingham, Alabama
  - Children's Hospital Orange County, Orange, California
  - University of California San Francisco, San Francisco, California
  - Helen De Vos, Grand Rapids, Michigan
  - New York Medical College, Valhalla, New York
  - Nationwide Children's Hospital, Columbus, Ohio

IPD SHARING:
Plan to Share IPD: No